CLINICAL TRIAL: NCT06642805
Title: Bilio-pancreatic Complications of Congenital Duodenal Obstructions
Acronym: Bilious
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC24_0157
Record Dates: First submitted 2024-10-04; First posted 2024-10-15 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Duodenal Obstruction
MeSH Terms: conditions — Duodenal Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort bilious
  Interventions: Procedure: duodenal atresia

INTERVENTIONS:
Procedure: duodenal atresia — surgery for duodenal atresia

SUMMARY:
Congenital duodenal obstructions, often grouped under the term duodenal atresias, encompass a range of malformations of the duodenum that cause partial or complete obstruction. In the long term, the main complications described fall within the spectrum of digestive occlusions (anastomotic stenosis, obstruction due to adhesions, and duodenal dysmotility) and may require surgical revisions. Biliary and pancreatic complications, which are embryologically logical, are reported in the form of rare clinical cases. The aim of the research is to identify biliopancreatic complications following duodenal atresia surgery in order to characterize them, estimate their national frequency, and determine any potential iatrogenic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery for duodenal atresia in a pediatric surgery department participating in the study over the past 20 years,
* legal representatives did not object to data collection

Exclusion Criteria:

* Patients ≥ 16 years at the time of surgery.
* Objection from the legal representatives of the child or the adult patient to the collection and use of health data

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients under 16 years who underwent surgery for duodenal atresia
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2028-12 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
frequency of biliar complication after surgical treatment of duodenal atresia | 1 year
frequency of pancreatic complication after surgical treatment of duodenal atresia | 1 year